CLINICAL TRIAL: NCT03313960
Title: A-One: A Randomized Controlled Trial Evaluating One Drop | Premium With Afrezza vs. One Drop | Premium Alone
Brief Title: A Randomized Controlled Trial Evaluating One Drop | Premium With Afrezza vs. One Drop | Premium Alone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Informed Data Systems, Inc. (Industry)
Collaborators: Mannkind Corporation (Industry)
Responsible Party: Principal Investigator, Chandra Osborn, PhD, MPH, Vice President, Health & Behavioral Informatics, Informed Data Systems, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-One
Record Dates: First submitted 2017-10-10; First posted 2017-10-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Afrezza
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- One Drop | Premium with Afrezza (Active Comparator)
  Interventions: Drug: Afrezza plus One Drop | Premium
- One Drop | Premium without Afrezza (Other)
  Interventions: Other: One Drop | Premium

INTERVENTIONS:
Drug: Afrezza plus One Drop | Premium — Participants in this group will receive insulin inhalation, prescribed by their physician, and will also receive One Drop | Premium (i.e., One Drop | Experts in-app coaching from a Certified Diabetes Educator (CDE) along with One Drop | Chrome Bluetooth-connected blood glucose meter that uploads results into the One Drop | Mobile app and 150 test strips per month for three months).
  Other Names: insulin inhalation
  Arms: One Drop | Premium with Afrezza
Other: One Drop | Premium — Participants in this group will receive One Drop | Premium (i.e., One Drop | Experts in-app CDE coaching with the One Drop | Chrome Bluetooth-connected blood glucose meter that uploads results into the One Drop | Mobile app and 150 test strips per month for three months).
  Arms: One Drop | Premium without Afrezza

SUMMARY:
The A-One study is a prospective, randomized controlled trial evaluating the use of the One Drop | Premium 'On Track' in combination with Afrezza treatment on the glycemic control, treatment adherence, social-cognitive barriers to adherence, and treatment satisfaction of people with Type 2 diabetes (T2D) and a hemoglobin A1c (A1c) > 7.0% already prescribed an injectable rapid-acting insulin.

DETAILED DESCRIPTION:
Eligible participants (N=400) with an A1c > 7.0% already prescribed a rapid-acting insulin will be randomized to one of two groups: (1) One Drop | Premium 'On Track' (i.e., use the One Drop | Mobile app with in-app diabetes education accredited by the American Diabetes Association with supplemental Afrezza content and a live Certified Diabetes Educator messaging in the app, the 'Chrome' Bluetooth-connected blood glucose meter that uploads blood glucose values in the app, and 150 test strips per month) in combination with Afrezza treatment (n=200) or (2) One Drop | Premium 'On Track' plus their current rapid-acting insulin (n=200).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Self-reported diagnosis of T2D
* Diagnosed with diabetes for at least 12 months
* Prescribed a prandial rapid-acting insulin
* Willing to take Afrezza rapid-acting insulin for 3 months instead of current rapid-acting insulin
* Willing to get a physician's prescription for Afrezza
* Self-reported A1c > 7.0% (later confirmed with a mail-in A1c laboratory test)
* Owns and uses an iPhone or Android phone with an operating system compatible with the One Drop | Mobile app
* Has successfully downloaded and used a smart phone application previously

Exclusion Criteria:

* Currently pregnant or planning to become pregnant during the trial period
* Cannot read or write in English
* Currently in a diabetes education or coaching program
* Had previously used One Drop | Premium or One Drop |
* Experts coaching
* Had previously used or is currently using Afrezza
* Currently smokes (cigaretts, e-cigs, pipes, cigars, marijuana) or has smoked anytime in the past 6 months
* Has chronic lung disease, e.g., COPD and asthma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months
  3-month between-group change in A1c assessed by a central lab

SECONDARY OUTCOMES:
Insulin Device Satisfaction | 3 months
  Within- and between-group change in insulin device satisfaction assessed by the Insulin Device Satisfaction Survey (IDSS)
Treatment Adherence | 3 months
  Within- and between-group change in treatment adherence assessed by the Adherence to Refills and Medications Scale for Diabetes (ARMS-D) and the Summary of Diabetes Self-care Activities Medications Subscale administered for each oral diabetes medication (SDSCA-MS) and insulin in the regimen (SDSCA-IS).
Self-care | 3 months
  Within- and between-group change in self-care assessed by the SDSCA's other subscales
Health-related Productivity | 3 months
  Within- and between-group change in health-related productivity assessed by the Work Productivity and Activity Impairment measure (WPAI).
Health-related Quality of Life | 3 months
  Within- and between-group change in health-related quality of life assessed by the Centers for Disease Control Health-related Quality of Life-14 (CDC HRQOL-14) and life satisfaction assessed by the Cantril Self-Anchoring Ladder of Life Satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Osborn, PhD, MPH, Principal Investigator — Informed Data Systems, Inc. | One Drop
Locations (1):
- One Drop, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Cramer JA. A systematic review of adherence with medications for diabetes. Diabetes Care. 2004 May;27(5):1218-24. doi: 10.2337/diacare.27.5.1218. PMID 15111553
- [Background] Davies MJ, Gagliardino JJ, Gray LJ, Khunti K, Mohan V, Hughes R. Real-world factors affecting adherence to insulin therapy in patients with Type 1 or Type 2 diabetes mellitus: a systematic review. Diabet Med. 2013 May;30(5):512-24. doi: 10.1111/dme.12128. PMID 23323988
- [Background] Feldman BS, Cohen-Stavi CJ, Leibowitz M, Hoshen MB, Singer SR, Bitterman H, Lieberman N, Balicer RD. Defining the role of medication adherence in poor glycemic control among a general adult population with diabetes. PLoS One. 2014 Sep 26;9(9):e108145. doi: 10.1371/journal.pone.0108145. eCollection 2014. PMID 25259843
- [Background] Piette JD, Wagner TH, Potter MB, Schillinger D. Health insurance status, cost-related medication underuse, and outcomes among diabetes patients in three systems of care. Med Care. 2004 Feb;42(2):102-9. doi: 10.1097/01.mlr.0000108742.26446.17. PMID 14734946
- [Background] Balkrishnan R, Rajagopalan R, Camacho FT, Huston SA, Murray FT, Anderson RT. Predictors of medication adherence and associated health care costs in an older population with type 2 diabetes mellitus: a longitudinal cohort study. Clin Ther. 2003 Nov;25(11):2958-71. doi: 10.1016/s0149-2918(03)80347-8. PMID 14693318
- [Background] Ho PM, Rumsfeld JS, Masoudi FA, McClure DL, Plomondon ME, Steiner JF, Magid DJ. Effect of medication nonadherence on hospitalization and mortality among patients with diabetes mellitus. Arch Intern Med. 2006 Sep 25;166(17):1836-41. doi: 10.1001/archinte.166.17.1836. PMID 17000939
- [Background] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Insulin adherence behaviours and barriers in the multinational Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabet Med. 2012 May;29(5):682-9. doi: 10.1111/j.1464-5491.2012.03605.x. PMID 22313123
- [Background] Lerman I, Diaz JP, Ibarguengoitia ME, Perez FJ, Villa AR, Velasco ML, Cruz RG, Rodrigo JA. Nonadherence to insulin therapy in low-income, type 2 diabetic patients. Endocr Pract. 2009 Jan-Feb;15(1):41-6. doi: 10.4158/EP.15.1.41. PMID 19211396
- [Background] Peyrot M, Rubin RR, Kruger DF, Travis LB. Correlates of insulin injection omission. Diabetes Care. 2010 Feb;33(2):240-5. doi: 10.2337/dc09-1348. PMID 20103556
- [Background] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Factors associated with injection omission/non-adherence in the Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabetes Obes Metab. 2012 Dec;14(12):1081-7. doi: 10.1111/j.1463-1326.2012.01636.x. Epub 2012 Jul 17. PMID 22726104
- [Background] Rubin RR, Peyrot M, Kruger DF, Travis LB. Barriers to insulin injection therapy: patient and health care provider perspectives. Diabetes Educ. 2009 Nov-Dec;35(6):1014-22. doi: 10.1177/0145721709345773. PMID 19934459
- [Background] Ross SA, Tildesley HD, Ashkenas J. Barriers to effective insulin treatment: the persistence of poor glycemic control in type 2 diabetes. Curr Med Res Opin. 2011 Nov;27 Suppl 3:13-20. doi: 10.1185/03007995.2011.621416. Epub 2011 Sep 23. PMID 21942467
- [Background] Baek RN, Tanenbaum ML, Gonzalez JS. Diabetes burden and diabetes distress: the buffering effect of social support. Ann Behav Med. 2014 Oct;48(2):145-55. doi: 10.1007/s12160-013-9585-4. PMID 24550072
- [Background] Gonzalez JS, Shreck E, Psaros C, Safren SA. Distress and type 2 diabetes-treatment adherence: A mediating role for perceived control. Health Psychol. 2015 May;34(5):505-13. doi: 10.1037/hea0000131. Epub 2014 Aug 11. PMID 25110840
- [Background] Nuffer W, Trujillo JM, Ellis SL. Technosphere insulin (Afrezza): a new, inhaled prandial insulin. Ann Pharmacother. 2015 Jan;49(1):99-106. doi: 10.1177/1060028014554648. Epub 2014 Oct 13. PMID 25313261
- [Background] Pittas AG, Westcott GP, Balk EM. Efficacy, safety, and patient acceptability of Technosphere inhaled insulin for people with diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2015 Nov;3(11):886-94. doi: 10.1016/S2213-8587(15)00280-6. Epub 2015 Sep 1. PMID 26341170
- [Background] Rosenstock J, Franco D, Korpachev V, Shumel B, Ma Y, Baughman R, Amin N, McGill JB; Affinity 2 Study Group. Inhaled Technosphere Insulin Versus Inhaled Technosphere Placebo in Insulin-Naive Subjects With Type 2 Diabetes Inadequately Controlled on Oral Antidiabetes Agents. Diabetes Care. 2015 Dec;38(12):2274-81. doi: 10.2337/dc15-0629. Epub 2015 Aug 7. PMID 26253730
- [Background] McPherson ML, Smith SW, Powers A, Zuckerman IH. Association between diabetes patients' knowledge about medications and their blood glucose control. Res Social Adm Pharm. 2008 Mar;4(1):37-45. doi: 10.1016/j.sapharm.2007.01.002. PMID 18342821
- [Background] Bradley C, Plowright R, Stewart J, Valentine J, Witthaus E. The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) evaluated in insulin glargine trials shows greater responsiveness to improvements than the original DTSQ. Health Qual Life Outcomes. 2007 Oct 10;5:57. doi: 10.1186/1477-7525-5-57. PMID 17927832
- [Background] Gonzalez JS, Schneider HE, Wexler DJ, Psaros C, Delahanty LM, Cagliero E, Safren SA. Validity of medication adherence self-reports in adults with type 2 diabetes. Diabetes Care. 2013 Apr;36(4):831-7. doi: 10.2337/dc12-0410. Epub 2012 Nov 30. PMID 23204245
- [Background] Mayberry LS, Gonzalez JS, Wallston KA, Kripalani S, Osborn CY. The ARMS-D out performs the SDSCA, but both are reliable, valid, and predict glycemic control. Diabetes Res Clin Pract. 2013 Nov;102(2):96-104. doi: 10.1016/j.diabres.2013.09.010. Epub 2013 Sep 26. PMID 24209600
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844